CLINICAL TRIAL: NCT05359666
Title: An Independent Review of Safety Data From a Closed Clinical Study Using Irrisept (Protocol IRR-CT-901-2013-01)
Brief Title: Retrospective Independent Safety Review of Closed Irrisept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLP-01
Record Dates: First submitted 2022-04-18; First posted 2022-05-04 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Adverse Events

STUDY DESIGN:
Intervention Model Description: The randomization methodology was controlled by the site for the IRR-CT-901-2013-01 trial. There was no additional randomization for CLP-01.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Irrisept (Experimental): Irrisept® was used for surgical irrigation in subjects with abdominal trauma or acute surgical abdomen for study protocol IRR-CT-901-2013-01.
  Interventions: Device: Irrisept
- Standard of Care (SoC) (Active Comparator): Institution determined the type of SoC used for surgical irrigation in subjects with abdominal trauma or acute surgical abdomen for study protocol IRR-CT-901-2013-01.
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Irrisept — Irrisept® is a manual, self-contained irrigation device designed for wound cleansing and irrigation. The solution is 0.05% Chlorhexidine Gluconate (CHG) in sterile water for irrigation, USP (99.95%). Irrisept contents include the solution, a 450 mL bottle, and the Irriprobe applicator. Irrisept is a manual, self-contained irrigation device that can produce 7-8 psi of pressure for effective wound cleansing and irrigation. The user squeezes the bottle to create streams of solution and directs the fluid from the applicator onto a wound. The mechanical action of the streams of fluid being applied over a wound removes particulates and debris.
  Subjects randomized to Irrisept on study protocol IRR-CT-901-2013-01 used the device, per the provided Instructions for Use. Those randomized to SoC received routine care, per the discretion of the investigator, and in accordance with the institution's guidelines.
  Arms: Irrisept
Device: Standard of Care — Subjects randomized to SoC on study protocol IRR-CT-901-2013-01 used any SoC type, per the investigator's discretion. SoC types were not standardized. Sites recorded SoC information as free text. The following were recorded as SoC types: Saline (recorded as "normal", "warm" and/or "sterile" saline or saline solution); Sodium Chloride (recorded as "sodium chloride (NACL)" or "NACL 0.9%"); "SoC"; Irrisept (recorded as "normal saline & Irrisept" and "Irrisept"); Chloraprep; "Gentamicin & saline"; unknown; and none.
  Arms: Standard of Care (SoC)

SUMMARY:
The purpose of CLP-01 was to complete the safety endpoint of the closed trial and ensure that all safety data generated by IRR-CT-901-2013-01 was accounted for and accurately identified, verified, and independently adjudicated. CLP-01 does not include an evaluation of the efficacy or exploratory endpoints from IRR-CT-901-2013-01. CLP-01 did not enroll new subjects and relied solely on data collected in the subject source and medical records in IRR-CT-901-2013-01. CLP-01 was conducted between March 2020 and November 2021.

DETAILED DESCRIPTION:
Between 2013 and 2016, Irrimax Corporation sponsored a prospective clinical study (IRR-CT-901-2013-01; NCT02255487) in the United States under IRB approval. IRR-CT-901-2013-01 defined primary and secondary efficacy, exploratory, and safety endpoints. The safety endpoint from IRR-CT-901-2013-01 was a clinical review and analysis of Adverse Events (AEs). However, IRR-CT-901-2013-01 was terminated early after the Interim Analysis primarily because of issues with the accuracy and completeness of the data collected for IRR-CT-901-2013-01, the lack of SoC standardization, and challenges assessing study endpoints arising out of the complexity of the trauma and co-morbidities of the subjects enrolled. The sole purpose of CLP-01 was to complete the safety endpoint for IRR-CT-901-2013-01.

CLP-01 reviewed all AEs recorded in IRR-CT-901-2013-01 and identified additional AEs in the subject source and medical records. All AEs were assessed for severity and causality and were reviewed by the individual Principal Investigators (PIs) at each site and the CLP-01 Medical Monitor (MM).

ELIGIBILITY:
Inclusion Criteria:

* Previously consented subjects from the closed study
* Subjects randomized to use Irrisept or SoC in the closed study
* Subjects who had a procedure in the hospital
* Subjects who used irrigation during the hospital procedure
* Subjects who had data that could be monitored and verified

Exclusion Criteria:

-Subjects who did not meet all inclusion criteria

The total number of subjects in this population - the mITT population - was 592.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chevy J Brown, MPH, Study Director — Director, Clinical Trials
Locations (17):
- United States (17):
  - University of Arizona Department of Surgery, Tucson, Arizona
  - Los Angeles County & USC Medical Center, Los Angeles, California
  - Denver Health Medical Center, Denver, Colorado
  - Tampa General Hospital University of South Florida (USF) College of Medicine, Tampa, Florida
  - University of Iowa Department of Surgery - 1504 JCP, Iowa City, Iowa
  - University of Kentucky Department of Surgery, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Baystate Medical Center Surgery Research, S3613, Springfield, Massachusetts
  - St. Louis University Department of Surgery, St Louis, Missouri
  - University of Cincinnati Division of Trauma/Critical Care Department of Surgery, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern (UTSW) Medical Center, Dallas, Texas
  - University of Texas Health Science Center (UTHSC) at Houston Center for Translational Injury Research, Houston, Texas
  - The University of Texas Health Center at San Antonio Division of Trauma and Emergency Surgery, San Antonio, Texas
  - University of Washington Harborview Medical Center Department of Surgery, Seattle, Washington
  - Medical College of Wisconsin Division of Trauma & Acute Care Surgery, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CLP-01, a retrospective review study conducted between 03/2020 & 11/2021, did not enroll new subjects, but relied solely on data collected for the trial IRR-CT-901-2013-01.CLP-01's purpose was to complete the safety endpoint of the closed trial & ensure that all safety data generated by IRR-CT-901-2013-01 was accounted for & accurately identified, verified, & independently adjudicated. CLP-01 did not include an evaluation of the efficacy or exploratory endpoints from IRR-CT-901-2013-01.
Pre-assignment Details: CLP-01 included safety data only from trial IRR-CT-901-2013-01. There were 636 ITT subjects (i.e., those who consented into IRR-CT-901-2013-01). There were 592 mITT subjects (i.e., those who consented, randomized to Irrisept or SoC, had a procedure, used irrigation during that procedure & had verifiable safety data. Of the 592 mITT subjects, 294 subjects were given Irrisept & 298 subjects were given SOC. The remaining 44 subjects had non-evaluable data & were not included in the analysis.
Groups:
- Irrisept: For subjects randomized to the investigational group, Irrisept was used during the surgical procedure, per the provided instructions for use.
  Irrisept® is a manual, self-contained irrigation device designed for wound cleansing and irrigation. The solution is 0.05% Chlorhexidine Gluconate (CHG) in sterile water for irrigation, USP (99.95%). Irrisept contents include the solution, a 450 mL bottle, and the Irriprobe applicator.
- Standard of Care (SoC): For subjects randomized to the control group, any SoC irrigation solution, preferred by the investigator, was used during the surgical procedure.
  SoC types were not standardized in IRR-CT-901-2013-01. The following were recorded as SoC types: Saline (recorded as "normal", "warm" and/or "sterile" saline or saline solution); Sodium Chloride (recorded as "sodium chloride (NACL)" or "NACL 0.9%"); "SoC"; Irrisept (recorded as "normal saline & Irrisept" and "Irrisept"); Chloroprep; "Gentamicin & saline"; unknown; and none.
Period: Overall Study
Arm/Group | Irrisept | Standard of Care (SoC)
Started | 294 (Of the 636 subjects within the ITT population, a total of 44 subjects had data that could not be verified. Their data was considered "non-evaluable" and excluded from the analysis. The randomization groups (i.e., Irrisept or SoC) for these 44 subjects could not be verified and is unknown. There were 294 subjects randomized to Irrisept in the mITT population.) | 298 (Of the 636 subjects within the ITT population, a total of 44 subjects had data that could not be verified. Their data was considered "non-evaluable" and excluded from the analysis. The randomization groups (i.e., Irrisept or SoC) for these 44 subjects could not be verified and is unknown. There were 298 subjects randomized to SoC in the mITT population.)
Completed | 294 | 298
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Although age, gender, race and/or region data was collected on the prior trial IRR-CT-901-2013-01, this information was not verified during CLP-01, as this was not the intent of the trial. The purpose of CLP-01 was to ensure safety data was accounted for and accurately identified, verified, and independently adjudicated. CLP-01 did not include an evaluation of the efficacy or exploratory endpoints from IRR-CT-901-2013-01.
Groups:
- Irrisept: For subjects randomized to the investigational group, Irrisept was used during the surgical procedure, per the provided instructions for use. Baseline data for age, gender, race and region was not the purpose of CLP-01 and therefore was not collected for Irrisept subjects. The purpose of CLP-01 was to identify and assess adverse event causality and severity only.
- Standard of Care (SoC): For subjects randomized to the control group, any SoC irrigation solution, preferred by the investigator, was used during the surgical procedure. Baseline data for age, gender, race and region was not the purpose of CLP-01 and therefore was not collected for SoC subjects. The purpose of CLP-01 was to identify and assess adverse event causality and severity only.
- Total: Total of all reporting groups
Arm/Group | Irrisept | Standard of Care (SoC) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: All Adverse Events
Description: The primary endpoint was identification of all adverse events from subjects that participated in the closed study (Protocol #IRR-CT-901-2013-01; NCT #02255487).
Time Frame: up to 30 +/- 3 days
Measure: Number; unit: Adverse Events
Groups:
- Irrisept: Irrisept® was used for surgical irrigation in subjects with abdominal trauma or acute surgical abdomen for study protocol IRR-CT-901-2013-01.
  Irrisept: Irrisept® is a manual, self-contained irrigation device designed for wound cleansing and irrigation. The solution is 0.05% Chlorhexidine Gluconate (CHG) in sterile water for irrigation, USP (99.95%). Irrisept contents include the solution, a 450 mL bottle, and the Irriprobe applicator. Irrisept is a manual, self-contained irrigation device that can produce 7-8 psi of pressure for effective wound cleansing and irrigation. The user squeezes the bottle to create streams of solution and directs the fluid from the applicator onto a wound. The mechanical action of the streams of fluid being applied over a wound removes particulates and debris.
  Subjects randomized to Irrisept on study protocol IRR-CT-901-2013-01 used the device, per the provided Instructions for Use.
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 294 | 298
Adverse Events | 894 | 962

2. Secondary Outcome: Subjects With Device-Related Adverse Events
Description: The secondary endpoint was identification of the number subjects with device-related adverse events from those that participated in the closed study (Protocol #IRR-CT-901-2013-01; NCT #02255487).
Time Frame: up to 30 +/- 3 days
Measure: Number; unit: Subjects with Device-related AEs
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 294 | 298
Subjects with Device-related AEs | 220 | 194

3. Secondary Outcome: Number of Device-Related Adverse Events
Description: Another secondary endpoint was identification of the overall number device-related adverse events from subjects that participated in the closed study (Protocol #IRR-CT-901-2013-01; NCT #02255487).
Time Frame: up to 30 +/- 3 days
Population: Of the total 1856 adverse events, 894 occurred in subjects on Irrisept and 962 occurred in subjects on SoC. There were 1808 total unrelated AEs (856 for Irrisept & 952 for SoC), 35 unlikely related AEs (30 for Irrisept & 5 for SoC), 13 possibly related AEs (8 for Irrisept & 5 for SoC) and 0 probably & definitely related AEs (0 for Irrisept & SoC).
Measure: Number; unit: Device-related AEs
Units Other Than Participants: Adverse Events
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 294 | 298
Number analyzed (Adverse Events) | 894 | 962
Device-related AEs
  Unrelated AEs | 856 | 952
  Unlikely Related AEs | 30 | 5
  Possibly Related AEs | 8 | 5
  Probably Related AEs | 0 | 0
  Definitely Related AEs | 0 | 0

4. Secondary Outcome: Number of Device Deficiencies
Description: For the Irrisept group only, any device deficiencies identified in the medical records and/or source documents (during the closed study when the study device was used, even if the deficiency was not associated with an AE), was recorded.
Time Frame: up to 30 +/- 3 days
Population: Device deficiencies were only reported for subjects randomized to Irrisept. Of the 294 subjects randomized to Irrisept, there were 43 device deficiencies. Device deficiencies were "any inadequacy of the medical device with respect to its identity, quality, durability, reliability, safety and/or performance".
Measure: Number; unit: Number of Device Deficiencies
Units Other Than Participants: Irrisept Device Deficiencies
Arm/Group | Irrisept
Number analyzed (Participants) | 294
Number analyzed (Irrisept Device Deficiencies) | 43
Number of Device Deficiencies
  Inadequate identification | 0
  Quality | 40
  Reliability | 0
  Safety | 0
  Performance | 0
  Malfunction | 0
  User Error | 3

ADVERSE EVENTS:
Time Frame: CLP-01 was a retrospective review study & did not enroll new subjects. AEs for subjects who participated in IRR-CT-901-2013-01 were reviewed beginning at informed consent completion, up to study completion (30 +/-3 days post-surgical procedure) or until AE resolution. CLP-01 relied solely on data collected in the subject source & medical records for the closed study in IRR-CT-901-2013-01. The study IRR-CT-901-2013-01 was conducted between 2015 and 2017.
Description: The following were collected: 1) # of SAEs, 2) all-cause mortality rates/randomization group & 3) categories of organ classes for all AEs & SAEs. No SADEs or USADEs were identified in CLP-01 for Irrisept or SoC. There was 1 ADE for 1 Irrisept subject; there were 0 SoC ADEs. All other AEs, anticipated or unanticipated, totaled 894 for Irrisept & 962 for SoC. There were 220 & 194 Irrisept & SoC subjects, respectively, that had AEs/SAEs/ADEs.
Arm/Group | Irrisept | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 7/294 | 8/298
Serious Adverse Events (participants affected / at risk) | 63/294 | 93/298
Other Adverse Events (participants affected / at risk) | 157/294 | 101/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irrisept (N=294) | Standard of Care (SoC) (N=298)
Blood/Lymphatic SAEs (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Cardiac SAEs (Cardiac disorders) | 5 (6) | 13 (15)
GI SAEs (Gastrointestinal disorders) | 17 (20) | 15 (16)
General SAEs (General disorders) | 2 (2) | 4 (4)
Hepatobiliary SAEs (Hepatobiliary disorders) | 1 (1) | 3 (3)
Infection SAEs (Infections and infestations) | 32 (37) | 29 (29)
Injury SAEs (Injury, poisoning and procedural complications) | 19 (22) | 19 (20)
Metabolic SAEs (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Nervous System SAEs (Nervous system disorders) | 5 (9) | 1 (2)
Psychiatric SAEs (Psychiatric disorders) | 0 (0) | 2 (2)
Renal/Urinary SAEs (Renal and urinary disorders) | 3 (3) | 3 (3)
Respiratory SAEs (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 16 (18)
Vascular SAEs (Vascular disorders) | 7 (7) | 6 (6)
Ear/Labyrinth SAEs (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Endocrine SAEs (Endocrine disorders) | 0 (0) | 0 (0)
Ocular SAEs (Eye disorders) | 0 (0) | 0 (0)
Immune System SAEs (Immune system disorders) | 0 (0) | 0 (0)
Investigational SAEs (Investigations) | 0 (0) | 0 (0)
Musculoskeletal SAEs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Neoplasm SAEs (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Reproductive System SAEs (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Skin/Subcutaneous Tissue SAEs (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irrisept (N=294) | Standard of Care (SoC) (N=298)
Blood/Lymphatic AEs (Blood and lymphatic system disorders) | 58 (101) | 60 (109)
Cardiac AEs (Cardiac disorders) | 48 (54) | 35 (37)
Ear/Labyrinth AEs (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine AEs (Endocrine disorders) | 3 (3) | 0 (0)
Ocular AEs (Eye disorders) | 1 (1) | 0 (0)
GI AEs (Gastrointestinal disorders) | 70 (98) | 74 (111)
General AEs (General disorders) | 39 (39) | 36 (37)
Hepatobiliary AEs (Hepatobiliary disorders) | 1 (1) | 4 (4)
Infection AEs (Infections and infestations) | 60 (67) | 52 (72)
Injury AEs (Injury, poisoning and procedural complications) | 51 (52) | 48 (50)
Investigational AEs (Investigations) | 5 (9) | 12 (15)
Metabolic AEs (Metabolism and nutrition disorders) | 62 (165) | 61 (192)
Musculoskeletal AEs (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
Neoplasm AEs (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Nervous System AEs (Nervous system disorders) | 9 (9) | 8 (10)
Psychiatric AEs (Psychiatric disorders) | 14 (17) | 17 (23)
Renal/Urinary AEs (Renal and urinary disorders) | 33 (34) | 30 (33)
Reproductive System AEs (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Respiratory AEs (Respiratory, thoracic and mediastinal disorders) | 47 (63) | 55 (76)
Skin/Subcutaneous Tissue AEs (Skin and subcutaneous tissue disorders) | 12 (12) | 16 (16)
Vascular AEs (Vascular disorders) | 29 (34) | 35 (44)
Adverse Device Effects (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT05359666/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05359666/SAP_001.pdf